CLINICAL TRIAL: NCT01290809
Title: Cognitive Sequelae of Prophylactic Cranial Irradiation in Non-small Cell Lung Cancer Patients
Brief Title: Prophylactic Cranial Irradiation (PCI) Cognitive Tests in Non-small Cell Lung Cancer (NSCLC) Patients
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: The Netherlands Cancer Institute (Other); Amsterdam UMC, location VUmc (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Maastricht University Medical Center (Other); University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 093074
Record Dates: First submitted 2011-02-01; First posted 2011-02-07 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: NSCLC
Keywords: Prophylactic Cranial Irradiation; lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Prophylactic Cranial Irradiation: NSCLC patients treated with whole brain PCI: cognitive functioning as assessed by neuropsychological tests?
- no Prophylactic Cranial Irradiation: NSCLC patients not treated with whole brain PCI: cognitive functioning as assessed by neuropsychological tests?

SUMMARY:
Stage III non-small cell lung cancer (NSCLC) patients constitute a significant proportion of the lung cancer population. The prognosis of these patients has improved over the years due the introduction of combined modality treatment, including high-dose chemo-radiotherapy. The brain, however, remains one of the major sites of failure. Patients with brain metastasis suffer from a variety of neurological, cognitive and emotional difficulties that are known to adversely affect the health-related quality of life. Prophylactic Cranial Irradiation (PCI) can prevent or delay the development of brain metastasis, and as such can improve neurological disease-free survival and consequently health-related quality of life. But survival is short, and toxicities are real, as PCI in itself can also induce adverse effects. The cognitive adverse effects of PCI are not sufficiently illuminated and documented, due to the lack of formal and systematic evaluation in patient populations expected to have short survival. Also, recent attempts to reduce cognitive side effects of PCI by the application of hippocampal-avoidance PCI in order to prevent memory deficits have not been fully evaluated yet.

Before PCI can be offered routinely to stage III NSCLC patients in daily practice, the costs and benefits of this therapy should be investigated properly, to allow for well-informed treatment choices.

ELIGIBILITY:
Inclusion Criteria:

* UICC stage III A or III B (without malignant pleural or pericardial effusion) non-small cell lung cancer
* Whole body PDG-PET scan before the start of therapy available: no distant metastasis.
* CT or preferably MRI of the brain before the start of radical therapy available; no brain metastasis.
* Platinum-based chemotherapy is mandatory.
* Radical local therapy: concurrent or sequential chemotherapy and radiotherapy with or without surgery.
* Radiotherapy dose without surgery to at least biological equivalent of 60 Gy.
* No prior cranial irradiation.sufficient proficiency in Dutch language
* sufficient proficiency in Dutch language
* MRI (and not CT scan) pre-PCI

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from 5 hospitals participating in the phase III trial: Prophylactic Cranial Irradiation (PCI) versus observation in radically treated patients with stage III non-small lung cancer: a phase III randomized study ((NVALT 11/DLCRG-02).
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2011-01; Primary Completion 2015-03 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
cognitive sequelae | 36 months
  The proposed study will investigate the cognitive sequelae of PCI in NSCLC patients in the context of a phase III randomized trial (Nederlandse vereniging van artsen voor longziekten en tuberculose: NVALT-11) on the efficacy of PCI in decreasing the proportion of NSCLC patients developing brain metastasis, and the impact of PCI on neurological symptoms and health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk deruysscher, Principal Investigator — Maastro Clinic, The Netherlands
Locations (4):
- Netherlands (4):
  - Academic Medical Center, Amsterdam
  - NKI, Amsterdam
  - VU University Medical Center, Amsterdam
  - University Medical Center Groningen, Groningen